CLINICAL TRIAL: NCT00573183
Title: Stimulant Abuser Groups to Engage in 12-Step (STAGE-12): Evaluation of a Combined Individual-Group Intervention to Reduce Stimulant and Other Drug Use by Increasing 12-Step Involvement
Brief Title: Stimulant Abuser Groups to Engage in 12-Step
Acronym: STAGE-12
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Dennis Donovan, Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIDA-CTN-0031; U10DA013714 (NIH)
Record Dates: First submitted 2007-12-13; First posted 2007-12-14 (Estimated); Results first posted 2014-01-29 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2016-10

CONDITIONS: Drug Abuse
Keywords: Cocaine, methamphetamine, amphetamine, other stimulant drugs
MeSH Terms: conditions — Substance-Related Disorders | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- STAGE-12 (Experimental): STAGE-12 received 3 individual and 5 group 12-step facilitation sessions focusing on 12-step principles plus an intensive referral in which counselors linked participants to community-based 12-step volunteers. These sessions took the place of 3 individual and 5 group sessions in the standard intensive outpatient drug treatment program and were integrated into treatment as usual.
  Interventions: Behavioral: STAGE-12
- Treatment as Usual (Active Comparator): Treatment as usual received standard care provided in intensive outpatient drug treatment program without the STAGE-12 components.
  Interventions: Behavioral: Treatment as Usual

INTERVENTIONS:
Behavioral: STAGE-12 — The STAGE-12 intervention will consist of a combination of five group and three individual sessions. The five group sessions will be taken from the Project MATCH Twelve Step Facilitation manual as modified for use with drug abusers and adapted for delivery in a group format. The group sessions will be augmented by three individual sessions derived from the introductory and termination sessions from the TSF manual and incorporating elements of the brief intensive 12-step referral procedure.
  Arms: STAGE-12
Behavioral: Treatment as Usual
  Arms: Treatment as Usual

SUMMARY:
The purpose of this study is to determine whether a combined group and individual 12-Step facilitative (TSF) intervention, Stimulant Abuser Groups to Engage in 12 -Step (STAGE-12), improves substance -related outcomes.

DETAILED DESCRIPTION:
This protocol is to evaluate the degree to which a combined group and individual 12-Step facilitative (TSF) intervention, Stimulant Abuser Groups to Engage in 12 -Step (STAGE-12), improves substance -related outcomes compared to treatment as usual (TAU) without STAGE-12 among stimulant abusers. The primary objective is to evaluate reduction in percent of days of stimulant use as measured by self-report. Secondary objectives include evaluating reduction in percent days of use of other substances, the degree to which STAGE-12 increases involvement in 12-step activities and attendance at 12-step meetings, and the extent to which such 12 -step involvement and meeting attendance mediate substance use outcomes.

ELIGIBILITY:
Inclusion Criteria:

* seeking outpatient treatment for stimulant abuse or dependence
* current diagnosis of stimulant abuse or dependence
* willing to participate in the protocol

Exclusion Criteria:

* not sufficiently medically or psychiatrically stable
* pending legal action that would inhibit their participation in the study
* in need of detoxification from opiates

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 471 (Actual)
Dates: Start 2008-01; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Donovan, Ph.D., Principal Investigator — University of Washington; Dennis Daley, Ph.D., Principal Investigator — Western Psychiatric Institute and Clinic
Locations (10):
- United States (10):
  - Gateway Community Services, Jacksonville, Florida
  - Hina Mauka Kaneohe Rehabilitation Services, Kaneohe, Hawaii
  - Maryhaven, Inc., Columbus, Ohio
  - Willamette Family Treatment Services, Eugene, Oregon
  - ChangePoint, Inc., Portland, Oregon
  - Addiction Medicine Services (WPIC), Pittsburgh, Pennsylvania
  - Dorchester Alcohol and Drug Commission, Summerville, South Carolina
  - Nexus Recovery Center, Dallas, Texas
  - Evergreen Manor, Inc., Everett, Washington
  - Recovery Centers of King County, Seattle, Washington

REFERENCES:
- [Result] Donovan DM, Daley DC, Brigham GS, Hodgkins CC, Perl HI, Garrett SB, Doyle SR, Floyd AS, Knox PC, Botero C, Kelly TM, Killeen TK, Hayes C, Kau'i Baumhofer N, Seamans C, Zammarelli L. Stimulant abuser groups to engage in 12-step: a multisite trial in the National Institute on Drug Abuse Clinical Trials Network. J Subst Abuse Treat. 2013 Jan;44(1):103-14. doi: 10.1016/j.jsat.2012.04.004. Epub 2012 May 31. PMID 22657748
- See also: Link to description of the STAGE-12 protocol on the NIDA Clinical Trials Network web site — http://www.drugabuse.gov/about-nida/organization/cctn/ctn/research-studies/stimulant-abuser-groups-to-engage-in-12-step-stage-12-evaluation-combined-i

RESULTS

PARTICIPANT FLOW:
Groups:
- STAGE-12: Received 3 individual and 5 group sessions focusing on 12-step principles plus an intensive referral in which counselors linked participants to community-based 12-step volunteers. These sessions took the place of 3 individual and 5 group sessions in the standard intensive outpatient drug treatment program.
- Treatment as Usual: Received standard care provided in intensive outpatient drug treatment program
Period: Overall Study
Arm/Group | STAGE-12 | Treatment as Usual
Started | 234 | 237
Completed | 162 | 174
Not Completed | 72 | 63
Not completed — Lost to Follow-up | 52 | 50
Not completed — Withdrawal by Subject | 8 | 2
Not completed — Death | 0 | 1
Not completed — Adverse Event | 2 | 0
Not completed — Incarceration | 5 | 8
Not completed — Other | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | STAGE-12 | Treatment as Usual | Total
Number analyzed (Participants) | 234 | 237 | 471
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 234 | 237 | 471
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.24 (10.04) | 38.45 (9.40) | 38.35 (9.71)
Gender [Count of Participants; unit: Participants]
  Female | 145 | 132 | 277
  Male | 89 | 105 | 194
Region of Enrollment [Number; unit: participants]
  United States | 234 | 237 | 471

OUTCOME MEASURES:

1. Primary Outcome: Days of Stimulant Use
Description: Number of days of use of stimulant drugs within 30-day blocks across a 6-month post-baseline period
Time Frame: 6 months
Population: The original sample size was based on power analysis and took attrition into account. Of the 471 individuals randomized to treatment, 50 subjects (TAU, n=20, STAGE-12, n=30) did not have any post-baseline measures and were therefore eliminated from the statistical analysis of the primary outcome and some of the secondary outcomes.
Measure: Mean (Standard Deviation); unit: days of stimulant use
Groups:
- Treatment as Usual: Standard treatment as usual in intensive outpatient substance abuse treatment program
- STAGE-12: Received 3 individual and 5 group sessions focusing on 12-step principles plus an intensive referral in which counselors linked participants to community-based 12-step volunteers. These sessions took the place of 3 individual and 5 group sessions.
Arm/Group | Treatment as Usual | STAGE-12
Number analyzed (Participants) | 217 | 204
days of stimulant use | 2.35 (5.39) | 2.13 (4.32)
Statistical Analysis 1: Comparison: Treatment as Usual vs STAGE-12; Mixture model with a logistic part for assessing zero-inflation and a negative binomial part for the over-dispersed count data, with corresponding 95% confidence intervals (CIs) of the odds ratios for logistic part and incidence rate ratios for negative binomial part; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis — 95% confidence interval; A covariate adjustment was used: average number of days of stimulant use within a 30-day window of assessment from 90 days pre-baseline to baseline; Odds Ratio (OR) = 3.3404, 95% CI 2-sided [1.2019 to 9.2842], Standard Error of Mean 0.4134 — The STAGE-12 group represented the numerator and TAU represented the reference group/denominator
Statistical Analysis 2: Comparison: Treatment as Usual vs STAGE-12; Test type: Superiority or Other; p < 0.01, Mixed Models Analysis; Odds Ratio (OR) = 2.4373, 95% CI 2-sided [1.0131 to 5.8637], Standard Error of Mean 0.4134

2. Secondary Outcome: Attendance at 12-step Meetings
Description: Days of attendance at 12-step meetings within 30-day blocks across a 6-month post-baseline period
Time Frame: 6 months
Population: The sample size was originally powered based on the primary outcome measure, not on the secondary 12-step measures.The analysis sample size was reduced due to missing values
Measure: Mean (Standard Deviation); unit: days of attending 12-step meetings
Arm/Group | STAGE-12 | Treatment as Usual
Number analyzed (Participants) | 189 | 206
days of attending 12-step meetings | 12.01 (9.73) | 10.52 (9.87)
Statistical Analysis 1: Comparison: STAGE-12 vs Treatment as Usual; Outcome measure: Number of days of self-reported Self-Help meeting attendance by the Substance Use Calendar (SUC) within a 30-day window of assessment at mid-treatment, end-of-treatment, first, second, third and last follow-ups; Test type: Superiority or Other; p < 0.05, Zero-inflated negative binomial random-e — Statistical Model - zero-inflated negative binomial random-effects regression; Statistical Model - zero-inflated negative binomial random-effects regression adjusted for average number of days of pre-baseline attendance

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | STAGE-12 | Treatment as Usual
Serious Adverse Events (participants affected / at risk) | 29/234 | 23/237
Other Adverse Events (participants affected / at risk) | 10/234 | 15/237
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | STAGE-12 (N=234) | Treatment as Usual (N=237)
angina pectoris (Cardiac disorders) | 1 (1) | 1 (1)
tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
GI haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
pancreatic cyst (Gastrointestinal disorders) | 1 (1) | 0 (0)
pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (2)
appendicitis (Infections and infestations) | 0 (0) | 1 (1)
catheter site infection (Infections and infestations) | 0 (0) | 1 (1)
cellulitis (Infections and infestations) | 1 (1) | 0 (0)
gateroenteritis viral (Infections and infestations) | 0 (0) | 1 (1)
hepatitis viral (Infections and infestations) | 0 (0) | 1 (1)
influenza (Infections and infestations) | 1 (1) | 0 (0)
pelvic inflamatory disease (Infections and infestations) | 0 (0) | 1 (1)
pneumonia (Infections and infestations) | 2 (3) | 1 (1)
pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0)
pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
sepsis (Infections and infestations) | 1 (1) | 0 (0)
stitch abscess (Infections and infestations) | 0 (0) | 1 (1)
viral infection (Infections and infestations) | 1 (1) | 0 (0)
accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
intentional overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
blood glucose increased (Investigations) | 1 (1) | 1 (1)
blood pressure increased (Investigations) | 1 (1) | 0 (0)
dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
coma (Nervous system disorders) | 1 (1) | 0 (0)
convulsion (Nervous system disorders) | 0 (0) | 1 (1)
partial seizure (Nervous system disorders) | 1 (1) | 0 (0)
syncope (Nervous system disorders) | 0 (0) | 1 (1)
anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
depression (Psychiatric disorders) | 3 (3) | 2 (2)
depression suicidal (Psychiatric disorders) | 1 (1) | 1 (1)
hallucination, auditory (Psychiatric disorders) | 0 (0) | 1 (1)
hallucination, mixed (Psychiatric disorders) | 0 (0) | 1 (1)
homicidal ideation (Psychiatric disorders) | 2 (2) | 0 (0)
suicidal ideation (Psychiatric disorders) | 6 (7) | 2 (2)
suicide attempt (Psychiatric disorders) | 3 (4) | 3 (4)
psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (1)
asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
rash papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
hypertension (Vascular disorders) | 0 (0) | 2 (2)
thrombosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | STAGE-12 (N=234) | Treatment as Usual (N=237)
pneumonia (Infections and infestations) | 7 (8) | 6 (7)
nasopharyngitis (Infections and infestations) | 4 (4) | 8 (9)
back pain (Musculoskeletal and connective tissue disorders) | 9 (9) | 5 (5)
depression (Psychiatric disorders) | 8 (8) | 8 (9)
suicidal ideation (Psychiatric disorders) | 10 (11) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes